CLINICAL TRIAL: NCT00068744
Title: Continuous Fluorouracil Plus Mitomycin C Versus Mitomycin C Plus Cisplatin As Chemotherapy Combination In Combined Radiochemotherapy For Locally Advanced Anal Cancer. A Phase II-III Study
Brief Title: Radiation Therapy, Mitomycin, and Either Fluorouracil or Cisplatin in Treating Patients With Locally Advanced Anal Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-22011-40014; EORTC-22011; EORTC-40014
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Anal Cancer
Keywords: squamous cell carcinoma of the anus; stage II anal cancer; stage IIIA anal cancer; stage IIIB anal cancer
MeSH Terms: conditions — Anus Neoplasms | interventions — Cisplatin; Fluorouracil; Mitomycin; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Drug: mitomycin C
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as mitomycin, fluorouracil, and cisplatin, use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells. It is not yet known whether radiation therapy and mitomycin are more effective when combined with fluorouracil or with cisplatin in treating anal cancer .

PURPOSE: This randomized phase II/III trial is studying how well giving radiation therapy and mitomycin together with fluorouracil works compared to radiation therapy, mitomycin, and cisplatin in treating patients with locally advanced anal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Phase II

* Primary

  * Compare the early clinical response (tumor response at 8 weeks) of patients with locally advanced anal cancer treated with radiotherapy with mitomycin and cisplatin vs mitomycin and fluorouracil.
* Secondary

  * Compare the feasibility of these regimens in these patients.
  * Compare the acute toxicity of these regimens in these patients.
  * Compare patient compliance to these regimens.

Phase III

* Primary

  * Compare the event-free survival of patients treated with these regimens.
* Secondary

  * Compare colostomy-free, disease-free, and overall survival of patients treated with these regimens.
  * Compare locoregional control in patients treated with these regimens.
  * Compare the late toxicity of these regimens in these patients.
  * Compare quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, T stage (T2 vs T3 vs T4), and nodal status (N0 vs N+). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy once daily 5 days a week on weeks 1-4, 7-8, and 3 days of week 9 (total of 33 fractions). Patients concurrently receive fluorouracil IV continuously on days 1-26 and 43-59 and mitomycin IV over 15 minutes on days 1 and 43.
* Arm II: Patients receive radiotherapy and mitomycin as in arm I and cisplatin IV over 1 hour on days 1, 8, 15, 22, 43, 50, and 57.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at weeks 12 and 26, and then every 6 months for 2 years.

Patients are followed every 2 weeks for 8 weeks, at week 26, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 678 patients (80 [40 per treatment arm] for phase II and 598 [299 per treatment arm] for phase III) will be accrued for this study within 2-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell anal carcinoma

  * Keratinizing or non-keratinizing
  * The following stages are eligible:

    * T2, N0, M0 with maximum tumor diameter at least 4 cm
    * T3-T4, N0, M0
    * Any T, N1-N3, M0
* Tumor located in the anal canal OR in the anal margin and infiltrating the anal canal
* No primary adenocarcinoma of the anus
* Measurable disease

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count greater than 2,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Not specified

Renal

* Creatinine less than 1.4 mg/dL

Cardiovascular

* No grade I angina pectoris with clinical symptoms within the past 3 months
* No grade II-IV angina pectoris within the past 3 months
* No stage II or greater distal arteritis

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy except adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No other concurrent radiotherapy

Surgery

* No prior colostomy

Other

* No prior treatment for anal cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2003-07; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Response as measured by RECIST at 8 weeks after completion of study treatment (Phase II)
Event-free survival as measured by Logrank at 12 and 26 weeks, then every 6 months thereafter (Phase III)

SECONDARY OUTCOMES:
Acute toxicity and compliance to treatment as measured by CTC v 2.0 at completion of study treatment (Phase II)
Colostomy-free survival as measured by Logrank at 12 and 26 weeks, then every 6 months thereafter (Phase III)
Overall survival as measured by Logrank at 12 and 26 weeks, then every 6 months thereafter
Disease-free survival as measured by Logrank at 12 and 26 weeks, then every 6 months thereafter
Local control as measured by Gray at 12 and 26 weeks, then every 6 months thereafter
Late toxicity as measured by RTOG and EROTC every 6 months after week 26
Quality of life as measured by EORTC Quality of Life Questionnaire-C30 and ASCT at 12 and 26 weeks, then every 6 months for 2 years after entry

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Bosset, MD, Study Chair — Hopital Jean Minjoz
Locations (24):
- Belgium (8):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Centre Hospitalier Lyon Sud, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Cazk Groeninghe - Campus Maria's Voorzienigheid, Kortrijk
  - U.Z. Gasthuisberg, Leuven
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
- National Cancer Institute of Egypt, Cairo, Egypt
- France (3):
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
- Germany (7):
  - Urologische Klinik - Universitaetsklinikum Aachen, Aachen
  - Charite - Campus Charite Mitte, Berlin
  - Robert Roessle Comprehensive Cancer Center - Charite Campus Buch, Berlin
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Halle, Halle
  - Onkologische Schwerpunktpraxis - Leer, Leer
  - Universitaetsklinikum Tuebingen, Tübingen
- Italy (2):
  - Ospedale Sant Anna, Como
  - Ospedale Busonera - Divisione Oncologia Medica, Padua
- Netherlands (2):
  - Arnhems Radiotherapeutisch Instituut, Arnhem
  - Dr. Bernard Verbeeten Instituut, Tilburg
- Institute of Oncology and Radiology of Serbia, Belgrade, Serbia

REFERENCES:
- [Result] Matzinger O, Roelofsen F, Mineur L, Koswig S, Van Der Steen-Banasik EM, Van Houtte P, Haustermans K, Radosevic-Jelic L, Mueller RP, Maingon P, Collette L, Bosset JF; EORTC Radiation Oncology and Gastrointestinal Tract Cancer Groups. Mitomycin C with continuous fluorouracil or with cisplatin in combination with radiotherapy for locally advanced anal cancer (European Organisation for Research and Treatment of Cancer phase II study 22011-40014). Eur J Cancer. 2009 Nov;45(16):2782-91. doi: 10.1016/j.ejca.2009.06.020. Epub 2009 Jul 28. PMID 19643599